CLINICAL TRIAL: NCT01724866
Title: Phase 2, Open-Label, Dose-Ranging Study of SPI-2012 (HM10460A) or Pegfilgrastim Use for the Management of Neutropenia in Patients With Breast Cancer Who Are Candidates for Adjuvant and Neoadjuvant Chemotherapy With the Docetaxel + Cyclophosphamide (TC) Regimen
Brief Title: Phase 2 Study of SPI-2012 or Pegfilgrastim for the Management of Neutropenia in Participants With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-GCF-12-201; 2013-003094-10 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-11-12 (Estimated); Results first posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-03

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia | interventions — eflapegrastim; pegfilgrastim; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: SPI-2012 45 µg/kg and Docetaxel + Cyclophosphamide (TC) (Experimental): Participants received SPI-2012 45 microgram/kilogram (µg/kg), subcutaneously (SC) once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 milligram/ square metre (mg/m^2) intravenous (IV) infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
  Interventions: Drug: SPI-2012; Drug: Docetaxel; Drug: Cyclophosphamide
- Arm 2: SPI-2012 135 µg/kg and Docetaxel + Cyclophosphamide (TC) (Experimental): Participants received SPI-2012 135 µg/kg, SC once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 mg/m^2 intravenous (IV) infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
  Interventions: Drug: SPI-2012; Drug: Docetaxel; Drug: Cyclophosphamide
- Arm 3: SPI-2012 270 µg/kg and Docetaxel + Cyclophosphamide (TC) (Experimental): Participants received SPI-2012 270 µg/kg, SC once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 mg/m^2 intravenous (IV) infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
  Interventions: Drug: SPI-2012; Drug: Docetaxel; Drug: Cyclophosphamide
- Arm 4: Pegfilgrastim and Docetaxel + Cyclophosphamide (TC) (Experimental): Participants received Pegfilgrastim 6 milligram (mg), SC once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 mg/m^2 intravenous (IV) infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
  Interventions: Drug: Pegfilgrastim; Drug: Docetaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: SPI-2012 — SPI-2012 SC injection.
  Other Names: Rolontis®; HM10460A; Eflapegrastim
  Arms: Arm 1: SPI-2012 45 µg/kg and Docetaxel + Cyclophosphamide (TC); Arm 2: SPI-2012 135 µg/kg and Docetaxel + Cyclophosphamide (TC); Arm 3: SPI-2012 270 µg/kg and Docetaxel + Cyclophosphamide (TC)
Drug: Pegfilgrastim — Pegfilgrastim SC injection, per manufacturer's Prescribing Information.
  Other Names: Neulasta®
  Arms: Arm 4: Pegfilgrastim and Docetaxel + Cyclophosphamide (TC)
Drug: Docetaxel — Docetaxel given based on standard dose for chemotherapy.
  Other Names: Taxotere
Drug: Cyclophosphamide — Cyclophosphamide given based on standard dose for chemotherapy.
  Other Names: Cytoxan

SUMMARY:
The purpose of this study is to assess the effect of test doses of SPI-2012 on the duration of severe neutropenia (DSN) during Cycle 1 in participants with breast cancer who are candidates for adjuvant or neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This is an open label, multicenter, dose ranging study, sequentially enrolled by study dose, with a non-inferiority design to compare the effectiveness of SPI-2012 relative to a fixed dose of pegfilgrastim as a concurrent active control to each dose of SPI-2012 in participants with breast cancer. This study included four arms comprising three dose levels of SPI-2012 (Arm 1: 45 µg/kg, Arm 2: 135 µg/kg, Arm 3: 270 µg/kg) versus pegfilgrastim (Arm 4: 6 mg). The start of study is defined as the initiation of treatment with SPI-2012 or pegfilgrastim. The duration of treatment consists of a maximum of 4 cycles (21 days per cycle) beginning on Day 1 with chemotherapy administration and continue through Day 21, plus a 30-day follow-up period, unless any of the discontinuation criteria applies.

The target population are participants with breast cancer who are candidates for neoadjuvant or adjuvant treatment with Docetaxel + Cyclophosphamide (TC) chemotherapy. All participants who receive at least 1 dose of either SPI-2012 or pegfilgrastim were followed for safety through 30 days after their last dose of study treatment or until all treatment-related adverse events (AEs) have resolved or returned to baseline/Grade 1, whichever is longer, or until it is determined that the outcome will not change with further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer and candidate for adjuvant or neoadjuvant chemotherapy
* Candidate for docetaxel and cyclophosphamide chemotherapy
* Female or male at least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Absolute neutrophil count (ANC) ≥ 1.5×109/L
* Platelet count ≥ 100 x 10^9/L
* Creatinine ≤ 1.5 x upper limit of normal (ULN)
* Total bilirubin ≤1.5 mg/dL(≤ 25.65 μmol/L).
* Aspartate aminotransferase per serum glutamic-oxaloacetic transaminase (AST/SGOT) and/or alanine aminotransferase per serum glutamic-pyruvic transaminase (ALT/SGPT) ≤ 2.5 x ULN
* Hemoglobin > 9 g/dL
* Alkaline phosphatase ≤ 1.5 x ULN

Exclusion Criteria:

* Known sensitivity to E. coli-derived products or known sensitivity to any of the products to be administered
* Known Human Immunodeficiency Virus (HIV) infection
* Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) diagnosis with detectable viral load or immunological evidence of chronic active disease
* Active infection or any serious underlying medical condition that would impair ability to receive protocol treatment
* Prior bone marrow or stem cell transplant
* Prolonged exposure to glucocorticosteroids and immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-03-25 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2014-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (10):
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Desert Springs Cancer Care, Scottsdale, Arizona
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Beaver Medical Group, Highland, California
  - California Cancer Associates for Research and Excellence, Los Angeles, California
  - Innovative Clinical Research Institute, Whittier, California
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - New York Oncology Hematology, PC, Albany, New York
  - North Shore Hematology/Oncology Associates, Setauket, New York
  - Good Samaritan Hospital, Corvallis, Corvallis, Oregon
- Australia (5):
  - Frankston Hospital, Frankston, Victoria
  - Royal Hobart, Brisbane
  - Ashford Cancer Center Research, Kurralta Park
  - Breast Cancer Research Center, WA, Perth
  - Ballarat Oncology & Haematology, Wendouree
- Georgia (2):
  - LTD " Cancer Center of Adjara Autonomic Republic", Batumi
  - Ltd ' Medulla - Chemotherapy and Immunotherapy Clinic, Tbilisi
- Hungary (5):
  - State Health Center, Budapest
  - National Institute of Oncology, Budapest
  - Uzsoki Hospital, Budapest
  - University Debrecen, Oncology Clinic, Debrecen
  - Szabolcs - Szatmár - Bereg megyei Kórházak és Egyetemi Oktatókórház, Nyíregyháza
- Ziv Medical Center, Safed, Israel
- Poland (4):
  - Regionalny Szpital Specjalistyczny, Grudziądz
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Dzienny Oddział Chemioterapii, Racibórz
  - MTZ Clinical Research Sp. z o.o., Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vacirca JL, Chan A, Mezei K, Adoo CS, Papai Z, McGregor K, Okera M, Horvath Z, Landherr L, Hanslik J, Hager SJ, Ibrahim EN, Rostom M, Bhat G, Choi MR, Reddy G, Tedesco KL, Agajanian R, Lang I, Schwartzberg LS. An open-label, dose-ranging study of Rolontis, a novel long-acting myeloid growth factor, in breast cancer. Cancer Med. 2018 May;7(5):1660-1669. doi: 10.1002/cam4.1388. Epub 2018 Mar 23. PMID 29573207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 27 investigative sites in the United States (10 sites), Australia (5 sites), Georgia (2 sites), Hungary (5 sites), Israel (1 site), and Poland (4 sites) from 25 March 2013 to 12 August 2014.
Pre-assignment Details: A total of 148 participants were randomized in the study, out of which 138 participants completed the study.
Groups:
- Arm 1: SPI-2012 45 µg/kg and Docetaxel + Cyclophosphamide (TC): Participants received SPI-2012 45 µg/kg, subcutaneously (SC) once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 mg/m^2 intravenous (IV) infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
- Arm 2: SPI-2012 135 µg/kg and TC: Participants received SPI-2012 135 µg/kg, SC once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 mg/m^2 IV infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
- Arm 3: SPI-2012 270 µg/kg and TC: Participants received SPI-2012 270 µg/kg, SC once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 mg/m^2 IV infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
- Arm 4: Pegfilgrastim and TC: Participants received Pegfilgrastim 6 mg, SC once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 mg/m^2 IV infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
Period: Overall Study
Arm/Group | Arm 1: SPI-2012 45 µg/kg and Docetaxel + Cyclophosphamide (TC) | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Started | 39 | 37 | 36 | 36
Evaluable Population (The Evaluable Population included all randomized participants who had received either SPI-2012 or pegfilgrastim and had completed Cycle 1.) | 39 | 36 | 36 | 36
Completed | 38 | 32 | 33 | 35
Not Completed | 1 | 5 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Initiation of Non-Protocol Therapy Either for Progressive Disease or Intolerance of TC Regimen | 0 | 2 | 0 | 0
Not completed — Investigator's Discretion | 0 | 1 | 1 | 0
Not completed — Need for Chemotherapy or Chemotherapy Regimen was Changed due to Amended HER2 Status | 1 | 0 | 0 | 0
Not completed — Participant Refused Further Treatment or Withdrew Consent | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Evaluable Population included all randomized participants who had received either SPI-2012 or pegfilgrastim and had completed Cycle 1.
Groups:
- Arm 1: SPI-2012 45 µg/kg and TC: Participants received SPI-2012 45 µg/kg, SC once per cycle on Day 2 of each cycle up to cycle 4 (each cycle was 21 days), approximately 24 hours after the administration of TC chemotherapy. TC chemotherapy was administered on Day 1 of each cycle as follows:
  Docetaxel 75 mg/m^2 IV infusion over 60 minutes and Cyclophosphamide 600 mg/m^2 IV infusion over 30-60 minutes.
- Total: Total of all reporting groups
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC | Total
Number analyzed (Participants) | 39 | 36 | 36 | 36 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.31) | 56.8 (10.63) | 55.7 (9.79) | 60.4 (10.43) | 58.2 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 34 | 36 | 144
  Male | 0 | 1 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 2 | 4 | 14
  Not Hispanic or Latino | 33 | 34 | 34 | 32 | 133
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 0 | 0 | 0 | 2
  White | 36 | 36 | 35 | 32 | 139
  Others | 0 | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Neutropenia (DSN) in Cycle 1
Description: DSN was defined as the interval from the day of first observation of severe neutropenia (ANC <0.5*10^9/L, Grade 4 neutropenia per NCI CTCAE) to the first ANC recovery to => 2.0*10^9/L in Cycle 1.
Time Frame: Cycle 1 (each cycle was 21 days)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 36 | 36 | 36
days | 1.03 (1.547) | 0.44 (1.275) | 0.03 (0.167) | 0.31 (0.822)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A 2-sided 95% confidence interval (CI) for the difference in mean DSN between any 2 arms was calculated. Non-inferiority p-value was calculated as two times the proportion of treatment difference greater than 1 in the resampling; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p = 0.296, Bootstrap method; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [0.19 to 1.27]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A 2-sided 95% CI for the difference in mean DSN between any 2 arms was calculated. Non-inferiority p-value was calculated as two times the proportion of treatment difference greater than 1 in the resampling; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p = 0.002, Bootstrap method; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.28 to 0.64]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A 2-sided 95% CI for the difference in mean DSN between any 2 arms was calculated. Non-inferiority p-values was calculated as two times the proportion of treatment difference greater than 1 in the resampling; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p < 0.001, Bootstrap method; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.56 to -0.06]

2. Secondary Outcome: Duration of DSN in Cycle 2
Description: DSN was defined as the interval from the day of first observation of severe neutropenia (ANC <0.5*10^9/L, Grade 4 neutropenia per NCI CTCAE) to the first ANC recovery to => 2.0*10^9/L in Cycle 2.
Time Frame: Cycle 2 (each cycle was 21 days)
Population: The Evaluable Population included all randomized participants who had received either SPI-2012 or pegfilgrastim and had completed Cycle 1. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 34 | 34 | 36
days | 0.46 (1.022) | 0.12 (0.478) | 0.03 (0.171) | 0.08 (0.368)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p = 0.001, Bootstrap method; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [0.06 to 0.74]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p < 0.001, Bootstrap method; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.16 to 0.24]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p < 0.001, Bootstrap method; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.19 to 0.06]

3. Secondary Outcome: Duration of DSN in Cycle 3
Description: DSN was defined as the interval from the day of first observation of severe neutropenia (ANC <0.5*10^9/L, Grade 4 neutropenia per NCI CTCAE) to the first ANC recovery to => 2.0*10^9/L in Cycle 3.
Time Frame: Cycle 3 (each cycle was 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 38 | 32 | 34 | 36
days | 0.45 (1.132) | 0.16 (0.628) | 0.15 (0.610) | 0.14 (0.593)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p = 0.002, Bootstrap method; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-0.07 to 0.72]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p < 0.001, Bootstrap method; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.27 to 0.30]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p < 0.001, Bootstrap method; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.27 to 0.28]

4. Secondary Outcome: Duration of DSN in Cycle 4
Description: DSN was defined as the interval from the day of first observation of severe neutropenia (ANC <0.5*10^9/L, Grade 4 neutropenia per NCI CTCAE) to the first ANC recovery to => 2.0*10^9/L in Cycle 4.
Time Frame: Cycle 4 (each cycle was 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 38 | 32 | 33 | 35
days | 1.05 (4.579) | 0.19 (0.738) | 0.09 (0.522) | 0.11 (0.404)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p = 0.781, Bootstrap method; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-0.01 to 2.47]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p < 0.001, Bootstrap method; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.17 to 0.38]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI was < 1 day; p < 0.001, Bootstrap method; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.23 to 0.22]

5. Secondary Outcome: Time to ANC Recovery in Cycle 1
Description: Time to ANC recovery was defined as the time from chemotherapy administration until ANC increased to ≥ 2×10^9/L after the expected nadir within Cycle 1. Time to ANC recovery was not calculated for participants whose ANC value didn't drop below 2 x10^9/L within Cycle 1.
Time Frame: Cycle 1 (each cycle was 21 days)
Population: The Evaluable Population included all randomized participants who had received either SPI-2012 or pegfilgrastim and had completed Cycle 1. Overall number of participants analyzed signifies the number of participants with recovery in Cycle 1.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 29 | 14 | 6 | 14
days | 10.0 [10.0 to 11.0] | 8.5 [8.0 to 9.0] | 8.0 [7.0 to 9.0] | 9.0 [8.0 to 10.0]
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.002, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [1.1 to 1.8]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.711, Log Rank; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.6 to 1.4]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.028, Log Rank; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.1 to 0.9]

6. Secondary Outcome: Time to ANC Recovery in Cycle 2
Description: Time to ANC recovery was defined as the time from chemotherapy administration until ANC increased to ≥2×10^9/L after the expected nadir within Cycle 2. Time to ANC recovery was not calculated for participants whose ANC value didn't drop below 2 x10^9/L within Cycle 2.
Time Frame: Cycle 2 (each cycle was 21 days)
Population: The Evaluable Population included all randomized participants who had received either SPI-2012 or pegfilgrastim and had completed Cycle 1. Overall number of participants analyzed signifies the number of participants with recovery in Cycle 2.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 23 | 8 | 7 | 10
days | 11.0 [10.0 to 11.0] | 9.5 [8.0 to 10.0] | 10.0 [8.0 to 14.0] | 10.0 [8.0 to 11.0]
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.672, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.8 to 1.4]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.348, Log Rank; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.5 to 1.3]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.973, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.4 to 2.9]

7. Secondary Outcome: Time to ANC Recovery in Cycle 3
Description: Time to ANC recovery was defined as the time from chemotherapy administration until ANC increased to ≥2×10^9/L after the expected nadir within Cycle 3. Time to ANC recovery was not calculated for participants whose ANC value didn't drop below 2 x10^9/L within Cycle 3.
Time Frame: Cycle 3 (each cycle was 21 days)
Population: The Evaluable Population included all randomized participants who had received either SPI-2012 or pegfilgrastim and had completed Cycle 1. Overall number of participants analyzed signifies the number of participants with recovery in Cycle 3.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 20 | 6 | 5 | 9
days | 10.0 [10.0 to 11.0] | 9.5 [8.0 to 12.0] | 9.0 [8.0 to 13.0] | 10.0 [9.0 to 11.0]
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.618, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.8 to 1.4]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.661, Log Rank; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.5 to 1.6]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.754, Log Rank; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.3 to 2.8]

8. Secondary Outcome: Time to ANC Recovery in Cycle 4
Description: Time to ANC recovery was defined as the time from chemotherapy administration until ANC increased to ≥2×10^9/L after the expected nadir within Cycle 4. Time to ANC recovery was not calculated for participants whose ANC value didn't drop below 2 x10^9/L within Cycle 4.
Time Frame: Cycle 4 (each cycle was 21 days)
Population: The Evaluable Population included all randomized participants who had received either SPI-2012 or pegfilgrastim and had completed Cycle 1. Overall number of participants analyzed signifies the number of participants with recovery in Cycle 4.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 23 | 8 | 4 | 12
days | 11.0 [10.0 to 13.0] | 10.0 [9.0 to 11.0] | 10.0 [8.0 to 14.0] | 10.0 [8.0 to 11.0]
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.009, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [1.1 to 1.7]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.527, Log Rank; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; A Cox proportional hazards model was used to estimate the hazard ratio and its two-sided 95% CI; Test type: Superiority; p = 0.815, Log Rank; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.4 to 3.9]

9. Secondary Outcome: Absolute Neutrophil Count (ANC) Nadir Overtime in Cycle 1
Description: Mean ANC nadir was defined as the mean of the lowest ANC value (*10^9/L) after administration of the study drug (SPI-2012 or pegfilgrastim) on any day in Days 1-3 of Cycle 1.
Time Frame: Cycle 1 (each cycle was 21 days)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 10^9 ANC per liter
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 36 | 36 | 36
10^9 ANC per liter | 1.5 (1.77) | 4.0 (3.86) | 7.2 (5.47) | 3.2 (2.43)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.008, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.911, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.002, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data

10. Secondary Outcome: Absolute ANC Nadir Overtime in Cycle 2
Description: Mean ANC nadir was defined as the mean of the lowest ANC value (*10^9/L) after administration of the study drug (SPI-2012 or pegfilgrastim) on any day in Days 1-3 of Cycle 2.
Time Frame: Cycle 2 (each cycle was 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 ANC/L
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 34 | 34 | 36
10^9 ANC/L | 2.0 (1.89) | 3.9 (2.55) | 6.8 (6.30) | 3.3 (2.16)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.005, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.633, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.027, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data

11. Secondary Outcome: Absolute ANC Nadir Overtime in Cycle 3
Description: Mean ANC nadir was defined as the mean of the lowest ANC value (*10^9/L) after administration of the study drug (SPI-2012 or pegfilgrastim) on any day in Days 1-3 of Cycle 3.
Time Frame: Cycle 3 (each cycle was 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 ANC/L
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 38 | 32 | 34 | 36
10^9 ANC/L | 2.3 (1.87) | 4.4 (3.26) | 6.1 (4.81) | 3.5 (1.92)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.015, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.571, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.066, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data

12. Secondary Outcome: Absolute ANC Nadir Overtime in Cycle 4
Description: Mean ANC nadir was defined as the mean of the lowest ANC value (*10^9/L) after administration of the study drug (SPI-2012 or pegfilgrastim) on any day in Days 1-3 of Cycle 4.
Time Frame: Cycle 4 (each cycle was 21 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 ANC/L
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 38 | 32 | 33 | 35
10^9 ANC/L | 2.1 (2.12) | 4.1 (2.86) | 4.8 (3.00) | 2.7 (1.64)
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.106, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.156, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.005, Asymptotic Normality Assumption; P-values was obtained based upon asymptotic normality assumption on the log10 transformed data

13. Secondary Outcome: Depth of ANC Nadir in Cycle 1
Description: Depth of ANC nadir was defined as the lowest Median ANC value (*10^9/L) after administration of the study drug (SPI-2012 or pegfilgrastim) on any day in Days 1-3 of Cycle 1.
Time Frame: Cycle 1 (each cycle was 21 days)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: 10^9 ANC/L
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 36 | 36 | 36
10^9 ANC/L | 0.8 [0.0 to 9.0] | 3.0 [0.1 to 14.1] | 6.2 [0.2 to 21.0] | 3.0 [0.0 to 9.1]
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 0.4, 95% CI 2-sided [0.25 to 0.80]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 1.0, 95% CI 2-sided [0.53 to 2.04]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 2.5, 95% CI 2-sided [1.40 to 4.54]

14. Secondary Outcome: Depth of ANC Nadir in Cycle 2
Description: Depth of ANC nadir was defined as the lowest Median ANC value (*10^9/L) after administration of the study drug (SPI-2012 or pegfilgrastim) on any day in Days 1-3 of Cycle 2.
Time Frame: Cycle 2 (each cycle was 21 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: 10^9 ANC/L
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 34 | 34 | 36
10^9 ANC/L | 1.3 [0.1 to 8.0] | 3.3 [0.1 to 9.5] | 4.8 [0.3 to 25.7] | 2.9 [0.1 to 9.2]
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 0.5, 95% CI 2-sided [0.30 to 0.80]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 1.1, 95% CI 2-sided [0.70 to 1.79]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 1.7, 95% CI 2-sided [1.07 to 2.79]

15. Secondary Outcome: Depth of ANC Nadir in Cycle 3
Description: Depth of ANC nadir was defined as the lowest Median ANC value (*10^9/L) after administration of the study drug (SPI-2012 or pegfilgrastim) on any day in Days 1-3 of Cycle 3.
Time Frame: Cycle 3 (each cycle was 21 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: 10^9 ANC/L
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 38 | 32 | 34 | 36
10^9 ANC/L | 1.9 [0.0 to 7.3] | 3.4 [0.1 to 12.3] | 4.1 [0.2 to 21.4] | 3.5 [0.1 to 8.1]
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 0.5, 95% CI 2-sided [0.34 to 0.89]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 1.1, 95% CI 2-sided [0.71 to 1.85]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 1.6, 95% CI 2-sided [0.97 to 2.49]

16. Secondary Outcome: Depth of ANC Nadir in Cycle 4
Description: Depth of ANC nadir was defined as the lowest Median ANC value (*10^9/L) after administration of the study drug (SPI-2012 or pegfilgrastim) on any day in Days 1-3 of Cycle 4.
Time Frame: Cycle 4 (each cycle was 21 days)
Population: as for outcome 2
Measure: Median (Full Range); unit: 10^9 ANC/L
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 38 | 32 | 33 | 35
10^9 ANC/L | 8.0 [0.0 to 9.2] | 4.2 [0.1 to 11.2] | 4.2 [0.4 to 11.9] | 2.4 [0.1 to 6.4]
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 0.7, 95% CI 2-sided [0.40 to 1.10]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 1.4, 95% CI 2-sided [0.87 to 2.38]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; Ratio = 1.9, 95% CI 2-sided [1.23 to 2.96]

17. Secondary Outcome: Time to ANC Nadir in Cycle 1
Description: Time to ANC nadir was defined as the time from chemotherapy administration until the occurrence of the ANC nadir.
Time Frame: Cycle 1 (each cycle was 21 days)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 36 | 36 | 36
Days | 8.0 [7.0 to 8.0] | 7.0 [7.0 to NA] — The upper limit of Kaplan-Meier 95% confidence interval was not estimable due to too many events at median value. | 7.0 [7.0 to 8.0] | 7.5 [7.0 to 16.0]

18. Secondary Outcome: Time to ANC Nadir in Cycle 2
Description: Time to ANC nadir was defined as the time from chemotherapy administration until the occurrence of the ANC nadir.
Time Frame: Cycle 2 (each cycle was 21 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 34 | 34 | 36
days | 8.0 [8.0 to NA] — The upper limit of Kaplan-Meier 95% confidence interval was not estimable due to too many events at median value. | 7.0 [7.0 to 8.0] | 8.0 [7.0 to 10.0] | 8.0 [7.0 to 15.0]

19. Secondary Outcome: Time to ANC Nadir in Cycle 3
Description: Time to ANC nadir was defined as the time from chemotherapy administration until the occurrence of the ANC nadir.
Time Frame: Cycle 3 (each cycle was 21 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 38 | 32 | 34 | 36
days | 8.0 [8.0 to NA] — The upper limit of Kaplan-Meier 95% confidence interval was not estimable due to too many events at median value. | 7.0 [7.0 to 8.0] | 8.0 [7.0 to 9.0] | 8.0 [7.0 to 15.0]

20. Secondary Outcome: Time to ANC Nadir in Cycle 4
Description: Time to ANC nadir was defined as the time from chemotherapy administration until the occurrence of the ANC nadir.
Time Frame: Cycle 4 (each cycle was 21 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 38 | 32 | 33 | 35
days | 8.0 [8.0 to NA] — The upper limit of Kaplan-Meier 95% confidence interval was not estimable due to too many events at median value. | 8.0 [7.0 to 8.0] | 8.0 [7.0 to 21.0] | 8.0 [7.0 to 8.0]

21. Secondary Outcome: Percentage of Participants With Febrile Neutropenia (FN) Across All Cycles From Cycle 1 to Cycle 4
Description: FN was defined as a temperature of more than 38.2 degree Celsius (°C) concurrent with an ANC greater than 0.5×10^9/L..
Time Frame: Cycle 1 to Cycle 4 (each cycle was 21 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 36 | 36 | 36
percentage of participants | 7.7 | 2.8 | 2.8 | 5.6
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 1.000, Fisher Exact; Percent Difference = 2.1, 95% CI 2-sided [-20.2 to 24.9]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 1.000, Fisher Exact; Percent Difference = -2.8, 95% CI 2-sided [-26.7 to 21.4]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 1.000, Fisher Exact; Percent Difference = -2.8, 95% CI 2-sided [-26.7 to 21.4]

22. Secondary Outcome: Number of Participants With Worst Grade Adverse Events (AEs), Deaths, Other Serious Adverse Events (SAEs), and Other AEs Leading to Discontinuation From Study Therapy, and Worst Grade Laboratory Abnormalities
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Participants with SAE other than death were reported.AE and Laboratory Abnormalities ("Hematology and Chemistry") were collected and graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03, where Grade 3 refers to severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated and Grade 4 refers to life-threatening consequences; urgent intervention indicated.
Time Frame: From the first dose up to 30 days post last dose of study drug (up to 4 months)
Population: The Safety Population included all randomized participants who had received at least one dose of any protocol specified drug (i.e., docetaxel, cyclophosphamide, SPI-2012 or pegfilgrastim).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 37 | 36 | 36
Participants
  Grade 3-4 TEAEs | 24 | 12 | 13 | 12
  Death | 0 | 0 | 0 | 0
  SAEs Other Than Death | 5 | 4 | 2 | 8
  TEAEs Leading to Discontinuation From Study Therapy | 0 | 2 | 1 | 1
  Grade 3-4 Lab Abnormalities: Hematology | 33 | 19 | 18 | 28
  Grade 3-4 Lab Abnormalities: Chemistry | 8 | 4 | 6 | 8

23. Secondary Outcome: Percentage of Participants With Hospitalization Across All Cycles From Cycle 1 to Cycle 4
Time Frame: All cycles from Cycle 1 to Cycle 4 (each cycle was 21 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
Number analyzed (Participants) | 39 | 36 | 36 | 36
percentage of participants | 7.7 | 8.3 | 2.8 | 13.9
Statistical Analysis 1: Comparison: Arm 1: SPI-2012 45 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.469, Fisher Exact; Percent Difference = -6.2, 95% CI 2-sided [-28.5 to 16.9]
Statistical Analysis 2: Comparison: Arm 2: SPI-2012 135 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.710, Fisher Exact; Percent Difference = -5.6, 95% CI 2-sided [-29.3 to 18.7]
Statistical Analysis 3: Comparison: Arm 3: SPI-2012 270 µg/kg and TC vs Arm 4: Pegfilgrastim and TC; Test type: Superiority; p = 0.199, Fisher Exact; Percent Difference = -11.1, 95% CI 2-sided [-34.6 to 13.3]

24. Secondary Outcome: Number of Participants With Positive Antibodies for SPI-2012
Description: Serum samples were to be tested in a screening assay for antibodies binding to SPI-2012 using a validated enzyme-linked immunosorbent assay (ELISA). Any serum samples positive for the antibody were to be tested in a confirmatory competitive inhibition assay using two antigens, SPI-2012 or granulocyte colony-stimulating factor (G-CSF), to confirm the presence of antibodies binding to SPI-2012 and to identify samples that were positive for antibodies binding to G-CSF.
Time Frame: Up to the end of the study (Approximately 3.5 months)
Population: The Evaluable Population included all randomized participants who had received either SPI-2012 or pegfilgrastim and had completed Cycle 1. Overall number of participants analyzed included participants who were treated with SPI-2012 and had post-treatment samples collected, and excluded participants who tested positive before being treated with SPI-2012. Data was collected and analyzed only for the "SPI-2012" reporting arms as per the planned analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC
Number analyzed (Participants) | 35 | 35 | 30
Participants | 0 | 0 | 2

25. Secondary Outcome: Time to Reach Maximum Concentration of SPI-2012 (Tmax)
Description: Blood samples were collected at specific time points to determine the serum concentrations of SPI-2012 and to derive pharmacokinetic (PK) parameters.
Time Frame: Pre-dose and at 1, 3, 6, 8, 10, 24, 48, 72, 144, 192, and 312 hours post-dose in Cycle 1 (each cycle was 21 days)
Population: The PK Population included subset of participants who had received at least one dose of SPI-2012 in Arms 1 to 3 and have sufficient number of blood samples. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: hours (hrs)
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC
Number analyzed (Participants) | 2 | 4 | 3
hours (hrs) | 58.7 [46.9 to 70.5] | 9.00 [8 to 48.1] | 24.0 [24 to 24.1]

26. Secondary Outcome: Maximum Concentration of SPI-2012 (Cmax)
Description: Blood samples were collected at specific time points to determine the serum concentrations of SPI-2012 and to derive PK parameters.
Time Frame: Pre-dose and at 1, 3, 6, 8, 10, 24, 48, 72, 144, 192, and 312 hours post-dose in Cycle 1 (each cycle was 21 days)
Population: The PK Population included subset of participants who had received at least one dose of SPI-2012 in Arms 1 to 3 and had sufficient number of blood samples. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC
Number analyzed (Participants) | 3 | 4 | 3
nanograms per milliliter (ng/mL) | 7.00 (6.08) | 247 (276) | 299 (329)

27. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to 312 Hours Post-Dose (AUC0-312)
Description: AUC(0-312) is the area under the serum concentration-time curve from time zero to 312 hour post dose calculated by the linear trapezoidal rule. Blood samples were collected at specific time points to determine the serum concentrations of SPI-2012 and to derive PK parameters.
Time Frame: Pre-dose and at 1, 3, 6, 8, 10, 24, 48, 72, 144, 192, and 312 hours post-dose in Cycle 1 (each cycle was 21 days)
Population: The PK Population included subset of participants who had received at least one dose of SPI-2012 in Arms 1 to 3 and have sufficient number of blood samples to estimate AUC. The AUC0-312 was not calculated for the 45 µg/kg dose due to insufficient data in the serum concentration profiles. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC
Number analyzed (Participants) | 0 | 2 | 3
nanogram*hour per milliliter (ng*hr/mL) |  | 16000 (5850) | 22900 (25100)

28. Secondary Outcome: Half-life of SPI-2012 (t1/2)
Description: t1/2 data were calculated and reported as harmonic mean and pseudo standard deviation (SD). Blood samples were collected at specific time points to determine the serum concentrations of SPI-2012 and to derive PK parameters.
Time Frame: Pre-dose and at 1, 3, 6, 8, 10, 24, 48, 72, 144, 192, and 312 hours post-dose in Cycle 1 (each cycle was 21 days)
Population: The PK Population included subset of participants who had received at least one dose of SPI-2012 in Arms 1 to 3 and had sufficient number of blood samples to estimate AUC. The t1/2 was not calculated for the 45 µg/kg arm because there were insufficient data in terminal phase of serum concentration profiles. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC
Number analyzed (Participants) | 0 | 2 | 1
hrs |  | 81.0 (88.4) | 31.5 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.

ADVERSE EVENTS:
Time Frame: From the first dose up to 30 days post last dose of study drug (up to 4 months)
Description: The Safety Population included all randomized participants who had received at least one dose of any protocol specified drug (i.e., docetaxel, cyclophosphamide, SPI-2012 or pegfilgrastim).
Arm/Group | Arm 1: SPI-2012 45 µg/kg and TC | Arm 2: SPI-2012 135 µg/kg and TC | Arm 3: SPI-2012 270 µg/kg and TC | Arm 4: Pegfilgrastim and TC
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 5/39 | 4/37 | 2/36 | 8/36
Other Adverse Events (participants affected / at risk) | 36/39 | 33/37 | 33/36 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: SPI-2012 45 µg/kg and TC (N=39) | Arm 2: SPI-2012 135 µg/kg and TC (N=37) | Arm 3: SPI-2012 270 µg/kg and TC (N=36) | Arm 4: Pegfilgrastim and TC (N=36)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 0
Gastritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: SPI-2012 45 µg/kg and TC (N=39) | Arm 2: SPI-2012 135 µg/kg and TC (N=37) | Arm 3: SPI-2012 270 µg/kg and TC (N=36) | Arm 4: Pegfilgrastim and TC (N=36)
Diarrhoea (Gastrointestinal disorders) | 17 | 7 | 14 | 15
Nausea (Gastrointestinal disorders) | 19 | 12 | 15 | 16
Asthenia (General disorders) | 5 | 2 | 5 | 8
Fatigue (General disorders) | 24 | 11 | 19 | 20
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 10 | 12 | 13
Headache (Nervous system disorders) | 12 | 5 | 8 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 18 | 12 | 13
Insomnia (Psychiatric disorders) | 3 | 5 | 5 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes